CLINICAL TRIAL: NCT03779282
Title: KETODEX for Emergence Delirium in Children Undergoing Outpatient Strabismus Surgery
Status: Completed | Type: Observational
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Khaled Dajani, Assistant Professor, Ochsner Health System
Other Study IDs: Pro00014439
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Emergence Delirium; Strabismus
MeSH Terms: conditions — Emergence Delirium; Strabismus | interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: pediatric patients undergoing outpatient strabismus surgery, and not receiving ketodex
- study: pediatric patients undergoing outpatient strabismus surgery, and receiving ketodex
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — see descriptions
  Other Names: ketamine
  Groups: study

SUMMARY:
Strabismus surgery for children is a very common procedure, with a high incidence of emergence delerium in the recovery room. A combination of intravenous ketamine/dexmedetomidine, or ketodex, has been previously shown to reduce emergence delerium in children undergoing adenotonsillectomy. Here, we study its application in strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II children undergoing outpatient strabismus surgery

Exclusion Criteria:

* anything not meeting the above

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy children, aged 0-18 years, undergoing outpatient strabismus surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium scale scores | up to 6 hours in recovery room
  A low total score would indicate less emergence delirium

SECONDARY OUTCOMES:
wong-baker or numeric pain scores, depending on age | up to 6 hours in recovery room
  A low total score would indicate less pain
discharge time | up to 24 hours
  time the patient is actually discharged from recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Dajani, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Main Campus, Jefferson, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hadi SM, Saleh AJ, Tang YZ, Daoud A, Mei X, Ouyang W. The effect of KETODEX on the incidence and severity of emergence agitation in children undergoing adenotonsillectomy using sevoflurane based-anesthesia. Int J Pediatr Otorhinolaryngol. 2015 May;79(5):671-6. doi: 10.1016/j.ijporl.2015.02.012. Epub 2015 Feb 19. PMID 25770644